CLINICAL TRIAL: NCT03108872
Title: Long Term Clinical Outcomes of Left Atrial Appendage Occlusion Versus New Oral Anticoagulants for Stroke Prevention in Patients With Non-valvular Atrial Fibrillation; From Korean Multicenter Registry
Brief Title: Left Atrial Appendage Occlusion Versus New Oral Anticoagulants for Stroke Prevention in Patients With Non-valvular Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sejong General Hospital (Other)
Collaborators: Korea University Anam Hospital (Other); Yonsei University (Other); Gachon University Gil Medical Center (Other); Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jong Lee, Principle Investigator, Sejong General Hospital
Other Study IDs: Ver 1.0_20170306
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation
Keywords: Anticoagulants; Atrial Appendage; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- LAAO group: One-hundred consecutive patients who underwent left atrial appendage occlusion from October 2010 to March 2015 in 5 Korean tertiary cardiovascular centers will be retrospectively registered.
  Interventions: Device: left atrial appendage occlusion
- NOAC group: Two-hundred age-, sex-, CHA2DS2-VASc score- and HAS-BLED score- matched control will be selected with a 1:2 ratio among all patients treated with new oral anticoagulants to prevent ischemic events from 5 centers during same periods
  Interventions: Drug: New oral anticoagulants

INTERVENTIONS:
Device: left atrial appendage occlusion — Percutaneous exclusion of left atrial appendage with Watchman or ACP devices
  Groups: LAAO group
Drug: New oral anticoagulants — Include dabigatran, rivaroxaban, apixaban and edoxaban
  Groups: NOAC group

SUMMARY:
We will compare long-term effectiveness and safety in patients with atrial fibrillation treated with left atrial appendage occlusion versus new oral anticoagulants to prevent ischemic stroke from multicenter registry data

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is associated with a substantial risk of stroke and systemic embolism. Vitamin K antagonists are highly effective in preventing stroke in patients with atrial fibrillation and high risk of ischemic stroke. However, their use is limited by a narrow therapeutic range, increased risk of intracranial hemorrhage, the need for continuous monitoring of INR, and drug or food interaction. New oral anticoagulants (NOACs), the direct thrombin inhibitor and the factor Xa inhibitor, have settled these limitations of warfarin therapy. In four pivotal phase 3 clinical trials and their meta-analysis, NOACs have been shown to significantly reduce ischemic stroke, intracranial hemorrhage, and mortality, and had similar major bleeding as for warfarin in patients with non-valvular atrial fibrillation (NVAF). Another new treatment strategy for prevention of stroke is left atrial appendage occlusion (LAAO). Left atrial appendage has been considered to be an origin of thrombi more than 90% of cases. The concept that exclusion of LAA from the circulation reduces the risk of stroke in patients with NVAF is therefore being tested in clinical studies. LAAO with Watchman device and only aspirin were proved to be non-inferior to warfarin for ischemic stroke prevention or systemic embolism. And, LAAO reduced significantly cardiac death and hemorrhagic stroke compared to warfarin in a long-term follow up. Up to date, there was no study to compare long-term clinical outcomes between LAAO and NOACs, which are two new treatment strategies for stroke prevention in patients with NVAF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrial fibrillation, who LAAO or NOAC to prevent ischemic stroke or systemic embolism
2. Patients with CHA2DS2-VASc score >1

Exclusion Criteria:

1. Patients who failed to successfully implant LAAO
2. Patients who receive new oral anticoagulant less than 6 months without clinical events
3. Patients with mitral stenosis more than mild grade
4. Patients with prosthetic heart valve

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation with high risk of ischemic stroke or systemic embolism
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness endpoint | During 4 years
  The composite of cardiovascular or unexplained death, or ischemic stroke, or systemic embolism
Primary safety endpoint | During 4 years
  Major bleeding or Serious device-related complications

SECONDARY OUTCOMES:
Cardiovascular or unexplained death | During 4 years
Ischemic stroke or systemic embolism | During 4 years
Hemorrhagic stroke | During 4 years
Major bleeding | During 4 years
  Bleeding event that required at least 2 units of packed RBCs or Symptomatic bleeding in a critical area or organ.
Serious device-related complications | During 4 years
  Serious pericardial effusion need procedure or surgery, peri-procedural stroke, or device embolization

CONTACTS AND LOCATIONS:
Locations (1):
- Sejong general hospital, 91-121 Sosa 2-Dong, Sosa-Gu, Bucheon-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Kim JS, Lee H, Suh Y, Pak HN, Hong GR, Shim CY, Yu CW, Lee HJ, Kang WC, Shin ES, Choi RK, Kar S, Park JW, Lim DS, Jang Y. Left Atrial Appendage Occlusion in Non-Valvular Atrial Fibrillation in a Korean Multi-Center Registry. Circ J. 2016 Apr 25;80(5):1123-30. doi: 10.1253/circj.CJ-15-1134. Epub 2016 Mar 17. PMID 26984716